CLINICAL TRIAL: NCT00035776
Title: Blood Factors and Peripheral Arterial Disease Outcomes
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1115; R01HL064739 (NIH)
Record Dates: First submitted 2002-05-04; First posted 2002-05-06 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2006-01

CONDITIONS: Arterial Occlusive Diseases; Cardiovascular Diseases; Peripheral Vascular Diseases; Coronary Disease
MeSH Terms: conditions — Arterial Occlusive Diseases; Cardiovascular Diseases; Peripheral Vascular Diseases; Coronary Disease

SUMMARY:
To investigate associations between hemostatic and inflammatory blood factors and progression of lower extremity arterial ischemia and cardiovascular events in men and women with and without lower extremity peripheral arterial disease.

DETAILED DESCRIPTION:
BACKGROUND:

The pathophysiology of functional impairment in patients with lower extremity peripheral arterial disease (PAD) is not well understood. Although lower ankle brachial index (ABI) levels are associated with greater functional impairment, one study suggests that the ABI improves to a greater degree than functional impairment after lower extremity revascularization. A meta-analysis of exercise studies in intermittent claudication demonstrated no significant association between improved walking ability after exercise and change in calf blood flow or ABI. Thus, characteristics in addition to ABI appear to influence walking ability in PAD.

It has been hypothesized that chronic inflammation is a biological mechanism underlying the decline in physical function that occurs with aging. It was recently reported that higher levels of D-dimer (fibrin degradation product) and high-sensitivity C-reactive protein (hsCRP) are associated with greater objectively assessed functional limitations in persons with PAD, but functional limitations refer to specific abilities, such as objectively measured walking speed or balance, which are distinct from disability. Furthermore, functional limitations may not fully explain disability.

DESIGN NARRATIVE:

The prospective study assessed associations between hemostatic and inflammatory blood factors and progression of lower extremity arterial ischemia and cardiovascular events in 346 men and women with lower extremity peripheral arterial disease (PAD) and 203 men and women without PAD.The study was ancillary to an NHLBI funded prospective study of functional and cardiovascular outcomes in men and women with PAD, the Walking and Leg Circulation Study (WALCS). The blood factors under study which included fibrinogen, PAI-1, TPA antigen, d-dimer, prothrombin 1.2, and C-reactive protein (CRP), were associated with progression of coronary atherosclerosis in proposed models of the pathogenesis of coronary atherosclerosis, but were not well studied in PAD.

There were two specific aims. The first was to determine whether higher baseline blood factor levels were associated with a) progression of lower extremity arterial ischemia (decline in ankle brachial index >= 0.15, lower extremity gangrene, ulcer, revascularization, or amputation); b) functional decline over a 48 month follow-up. The second aim was to determine whether higher baseline blood factor levels were associated with new cardiovascular events over a 48 month follow-up. The hypothesis was that higher blood factor levels at baseline would be associated with PAD progression, functional decline, and higher rates of cardiovascular morbidity and mortality

Pilot data from the Cardiovascular Health Study (CHS) showed that relative risks of fibrinogen, D-dimer and CRP levels for cardiovascular events were highest for events occurring more proximate to baseline blood factor measurements. Therefore, the study also sought to determine whether blood factor levels measured at the most recent examination prior to cardiovascular events or PAD progression were higher than the levels that did not immediately precede cardiovascular events or PAD progression. The hypothesis was tested that blood factor levels at the most recent examination prior to cardiovascular events or PAD progression would be higher than blood factor levels that did not immediately precede cardiovascular events.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-01; Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary McDermott — Northwestern University

REFERENCES:
- [Background] McDermott MM, Guralnik JM, Greenland P, Pearce WH, Criqui MH, Liu K, Taylor L, Chan C, Sharma L, Schneider JR, Ridker PM, Green D, Quann M. Statin use and leg functioning in patients with and without lower-extremity peripheral arterial disease. Circulation. 2003 Feb 11;107(5):757-61. doi: 10.1161/01.cir.0000050380.64025.07. PMID 12578881
- [Background] McDermott MM, Green D, Greenland P, Liu K, Criqui MH, Chan C, Guralnik JM, Pearce WH, Ridker PM, Taylor L, Rifai N, Schneider JR. Relation of levels of hemostatic factors and inflammatory markers to the ankle brachial index. Am J Cardiol. 2003 Jul 15;92(2):194-9. doi: 10.1016/s0002-9149(03)00537-x. PMID 12860223
- [Background] McDermott MM, Greenland P, Green D, Guralnik JM, Criqui MH, Liu K, Chan C, Pearce WH, Taylor L, Ridker PM, Schneider JR, Martin G, Rifai N, Quann M, Fornage M. D-dimer, inflammatory markers, and lower extremity functioning in patients with and without peripheral arterial disease. Circulation. 2003 Jul 1;107(25):3191-8. doi: 10.1161/01.CIR.0000074227.53616.CC. Epub 2003 Jun 16. PMID 12810614
- [Background] McDermott MM, Guralnik JM, Greenland P, Green D, Liu K, Ridker PM, Chan C, Criqui MH, Ferrucci L, Taylor LM, Pearce WH, Schneider JR, Oskin SI. Inflammatory and thrombotic blood markers and walking-related disability in men and women with and without peripheral arterial disease. J Am Geriatr Soc. 2004 Nov;52(11):1888-94. doi: 10.1111/j.1532-5415.2004.52514.x. PMID 15507067
- [Background] McDermott MM, Greenland P, Guralnik JM, Ferrucci L, Green D, Liu K, Criqui MH, Schneider JR, Chan C, Ridker P, Pearce WH, Martin G, Clark E, Taylor L. Inflammatory markers, D-dimer, pro-thrombotic factors, and physical activity levels in patients with peripheral arterial disease. Vasc Med. 2004 May;9(2):107-15. doi: 10.1191/1358863x04vm525oa. PMID 15521700
- [Background] Shadman R, Criqui MH, Bundens WP, Fronek A, Denenberg JO, Gamst AC, McDermott MM. Subclavian artery stenosis: prevalence, risk factors, and association with cardiovascular diseases. J Am Coll Cardiol. 2004 Aug 4;44(3):618-23. doi: 10.1016/j.jacc.2004.04.044. PMID 15358030
- [Background] McDermott MM, Liu K, Greenland P, Guralnik JM, Criqui MH, Chan C, Pearce WH, Schneider JR, Ferrucci L, Celic L, Taylor LM, Vonesh E, Martin GJ, Clark E. Functional decline in peripheral arterial disease: associations with the ankle brachial index and leg symptoms. JAMA. 2004 Jul 28;292(4):453-61. doi: 10.1001/jama.292.4.453. PMID 15280343
- [Background] McDermott MM, Liu K, Ferrucci L, Criqui MH, Greenland P, Guralnik JM, Tian L, Schneider JR, Pearce WH, Tan J, Martin GJ. Physical performance in peripheral arterial disease: a slower rate of decline in patients who walk more. Ann Intern Med. 2006 Jan 3;144(1):10-20. doi: 10.7326/0003-4819-144-1-200601030-00005. PMID 16389250
- [Background] McDermott MM, Guralnik JM, Ferrucci L, Criqui MH, Greenland P, Tian L, Liu K, Tan J. Functional decline in lower-extremity peripheral arterial disease: associations with comorbidity, gender, and race. J Vasc Surg. 2005 Dec;42(6):1131-7. doi: 10.1016/j.jvs.2005.08.010. PMID 16376203
- [Background] McDermott MM, Ferrucci L, Liu K, Criqui MH, Greenland P, Green D, Guralnik JM, Ridker PM, Taylor LM, Rifai N, Tian L, Zheng J, Pearce WH, Schneider JR, Vonesh E. D-dimer and inflammatory markers as predictors of functional decline in men and women with and without peripheral arterial disease. J Am Geriatr Soc. 2005 Oct;53(10):1688-96. doi: 10.1111/j.1532-5415.2005.53510.x. PMID 16181167